CLINICAL TRIAL: NCT02245113
Title: Effects of High Oleic Palm Olein (HOPO), Virgin Olive Oil (OO) and Refined Bleached and Deodorized (RBD) Coconut Oil (CO) Diets on Lipid Profile, Markers of Insulin Resistance, Inflammatory and Obesity in Overweight Subject.
Brief Title: Effects of High Oleic Palm Olein, Virgin Olive Oil and Coconut Oil Diets on Markers Selected in Malaysian
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Universiti Putra Malaysia (Other); IMU University, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: R002302000
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test Fat P (Experimental): Test fat, n= 10 (minimum), 6 weeks intervention, Intervention 1, Intervention 2, and Intervention 3.
  Interventions: Other: diets
- Test Fat Q (Experimental): Test fat, n= 10 (minimum), 6 weeks intervention, Intervention 1, Intervention 2, and Intervention 3.
  Interventions: Other: diets
- Test Fat R (Experimental): Test fat, n= 10 (minimum), 6 weeks intervention, Intervention 1, Intervention 2, and Intervention 3.
  Interventions: Other: diets

INTERVENTIONS:
Other: diets — Feeding trial for 6 weeks (week 0 - baseline). The experimental diets are comprised of 30% kcal fat, 15% kcal protein and 55% kcal carbohydrate. Each of the test fat contributes to two-thirds of total dietary fat will be compared.

SUMMARY:
This study will be comparing human body responses by the effects of diets cooked with NoveLin, virgin olive oil and RBD coconut oil.

DETAILED DESCRIPTION:
NoveLin has high content of monounsaturate fatty acids - oleic acid (C18:1) which is the predominant fatty acid and in this study NoveLin is used as cooking fat in compare with olive oil. Olive oil is the world's most commonly eaten monounsaturated oil which contains 55 - 83% oleic acid. Consumption of olive oil gives numerous health benefits on lowering total and LDL cholesterol, reducing LDL cholesterol's, lowering blood clotting factors, and lowering blood pressure. Coconut oil is the richest source of medium chain fatty acid and it has greater than 90% of saturated fatty acid with dominant fatty acid of lauric acid (C12:0). RBD coconut oil is used as positive control in this study.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 20-60 years
* BMI 23 - 27.5 kg/m2
* free from any disease
* not on any medication or treatment associated with reduction of CVD
* non-smokers and non-heavy drinker or having smoking or alcoholic history
* not pregnant or lactating
* willing and able to comply

Exclusion Criteria:

* people on weight reduction therapy/program
* people on cholesterol reduction medicatio
* have one or more of the chronic diseases
* people with blood clotting problem/ coagulopathy / deep vein thrombosis.
* hypertensive persons (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg)
* female who is pregnant
* people travel to overseas during feeding.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
change in c-peptide level | week 0(baseline) and week 6

SECONDARY OUTCOMES:
change in insulin resistance's markers | week 0(baseline) and week 6
change in inflammatory markers | week 0(baseline) and week 6
change in obesity markers | week 0(baseline) and week 6
change in lipid profile | week 0(baseline) and week 6
change in physical characteristic (eg. BMI, body weight) | week 0(baseline) and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Voon Phooi Tee, PhD, Principal Investigator — MPOB; Lee Sin Tien, BSc, Principal Investigator — UPM; Norhaizan Md Esa, PhD, Principal Investigator — UPM; Tony Ng Kock Wai, PhD, Principal Investigator — IMU; Verna Lee Kar Mun, PhD, Principal Investigator — IMU
Locations (1):
- MPOB, Kajang, Selangor, Malaysia